CLINICAL TRIAL: NCT01472211
Title: An Efficacy Trial of a Gravity-fed Household Water Treatment Device as a Delivery System for Zinc in Zinc Deficient Preschool Children and Pregnant Women From Rural Settings With Poor Access to Potable Water in Benin.
Brief Title: Water-based Zinc Intervention Trial in Zinc Deficient Children
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Zn released from vehicle led to fortification levels higher than planned. New filter will be developed.
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Université d'Abomey-Calavi (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSF_zinc_study
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Zinc Deficiency; Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Disinfection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- intervention filter (Experimental): children consuming purified and zinc enriched water delivered by a household-based water filter
  Interventions: Device: zinc enriching filter (LifeStrawFamily)
- placebo filter (Placebo Comparator): children consuming purified water delivered by a household-based water filter
  Interventions: Device: placebo filter
- disinfection tablets (Active Comparator): children will consume water treated with government promoted disinfection tablets (aquatabs)
  Interventions: Other: disinfection tablets

INTERVENTIONS:
Device: zinc enriching filter (LifeStrawFamily) — filter purifies water and enriches it with zinc at 1-4 mg/l.
  Other Names: LifeStrawFamily by Vestergaards-Frandsen (Switzerland)
  Arms: intervention filter
Device: placebo filter — filter purifies water
  Other Names: LifeStrawFamily by Vestergaards-Frandsen (Switzerland)
  Arms: placebo filter
Other: disinfection tablets — government promoted tablets disinfect water
  Other Names: Aquatabs water purification tablets
  Arms: disinfection tablets

SUMMARY:
The overall aim of this trial is to determine whether the use of the household-based water treatment device Life Straw Family (LSF) can be an effective strategy to improve zinc status and health status of vulnerable populations in developing country rural settings with poor access to potable water.

To assess the effectiveness of the LSF strategy (a filter delivering purified and zinc enriched water) a double blind controlled field efficacy trial will take place over a period of 12 months in rural villages in the district of Natitingou, North-West Benin. In order to attain the research objectives the efficacy trial will envisage 3 arms: intervention (zinc enriching filter), placebo (filter) and control group (disinfection tables). During the trial the following outcomes will be monitored: zinc status and growth rate of the participating children, zinc status and pregnancy outcome in a sub-sample of pregnant women (pregnancy sub-study), diarrhea prevalence in all participating subjects, water quality, zinc enrichment of water, and modality and consistency of use of the LSF-device by the study population.

The study hypotheses are: 1) the use of the LSF-device will reduce microbiological contamination of the household water, 2) the use of the LSF-device will increase zinc intakes and serum zinc concentration in preschool children, 3) the use of the LSF-device will increase zinc intakes and serum zinc concentration in pregnant women, 4) the achievement of 1 and 2 will improve growth and lower frequency and length of diarrhea episodes in participating preschool children, 5) the achievement of 1 and 3 will improve pregnancy outcome and lower frequency and length of diarrhea episodes in participating pregnant women, 6) the use of the LSF-device will lower frequency and length of diarrhea episodes in participating households members.

ELIGIBILITY:
Inclusion Criteria:

* 2-5 year old children
* subjects residing in the study area for the whole study period

Exclusion Criteria:

* subject with severe anemia (Hb < 7 g/dl)
* subjects affected by chronic medical illnesses known to interact with zinc metabolism
* subjects receiving zinc supplementation or other medicines that may affect zinc metabolism

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 317 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Zinc status | 12 months
  At baseline, endpoint and at a randomly assigned screening between month 1 and 11, a 6 ml whole blood sample will be collected by venipuncture in 2-5y children (N=270). The blood sample will be used to determine concentration of zinc in the serum (SZn). Inflammation indicator C-reactive protein (CRP) will be analysed to adjust SZn values.

SECONDARY OUTCOMES:
Gut microbiota characterisation | 2 months
  At baseline and month 2, stool samples will be collected in 60 children (20 per study arm) for gut flora characterisation.
Iron status | 12 months
  At baseline, endpoint and at a randomly assigned screening between month 1 and 11, a 6 ml whole blood sample will be collected by venipuncture in 2-5y children (N=270). The blood sample will be used to determine the levels of haemoglobin (Hb) and serum ferritin (SF) for the assessment of iron status.
Growth rate | 12 months
  At baseline, midpoint and endpoint weight, height and MUAC will be measured in 2-5y children (N=270). Anthropometric measurements will be used to determine growth rate.
Diarrhea prevalence | 12 months
  Study children will be weekly surveyed for diarrhea occurrence. Mothers/tutors will be requested to report any diarrhea episode occurred in the last 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof. Dr.med., Study Chair — Swiss Federal Institute of Technology
Locations (1):
- Hopital de Zone, Natitingou, Atakora Department, Benin

REFERENCES:
- [Derived] Galetti V, Mitchikpe CE, Kujinga P, Tossou F, Hounhouigan DJ, Zimmermann MB, Moretti D. Rural Beninese Children Are at Risk of Zinc Deficiency According to Stunting Prevalence and Plasma Zinc Concentration but Not Dietary Zinc Intakes. J Nutr. 2016 Jan;146(1):114-23. doi: 10.3945/jn.115.216606. Epub 2015 Nov 25. PMID 26609168